CLINICAL TRIAL: NCT04770129
Title: Demographic Data and Outcomes Of Metastatic Breast Cancer Patients Treated Over The Last Decade At Tertiary Oncology Clinics In Highly Populated Cities In Turkey: A Turkish Oncology Collaborative Group Analysis
Brief Title: Real-World Data on Clinical Characteristics, Demographics, and Outcomes of Patients With Metastatic Breast Cancer in Turkey
Status: Completed | Type: Observational
Sponsor: Turkish Oncology Group (Network)
Collaborators: Acibadem Maslak Hospital (Other); Ege University Hospital (Unknown); Marmara University Pendik Training and Research Hospital (Other); Acibadem Altunizade Hospital, Istanbul (Unknown); Istanbul University (Other); V.K.V. American Hospital, Istanbul (Other); Hacettepe University (Other)
Responsible Party: Principal Investigator, Yesim Eralp, Prof. Dr., Acibadem Maslak Hospital
Other Study IDs: ML42450
Record Dates: First submitted 2021-02-15; First posted 2021-02-25 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time period 2010-2014: Data from Turkish participants with metastatic breast cancer diagnosed January 2010-December 2014 will be retrospectively collected.
- Time period 2015-2019: Data from Turkish participants with metastatic breast cancer diagnosed January 2015-December 2019 will be retrospectively collected.

SUMMARY:
This study is planned as a secondary data use (SDU) study and the data collection will be performed retrospectively. Patients who presented to the participating sites with metastatic breast cancer will be defined, and patients' data will be recorded into a database.

DETAILED DESCRIPTION:
This study is planned as a secondary data use (SDU) study and the data collection will be performed retrospectively. Patients who presented to the participating sites with metastatic breast cancer will be defined and patients' data will be recorded into a database. The study will be performed at clinical centers located in the populated cities with high clinical and diagnostic standards including patients presented with metastatic disease will be recorded. It is also planned to collect data on the treatment of metastatic breast cancer in line with institutional guidelines at academic and private centers which has implemented high quality clinical and pathologic standards.

This retrospective study is designed to record, define and evaluate the changes in the presentation patterns, pathological subtypes and outcomes of metastatic breast cancer patients in relation with the evolution of overall and progression-free survival rates following the changes in treatment approaches over the last decade based on the evolving/different treatment regimens of metastatic breast cancer.

These findings will shed light on how changes in metastatic patterns have influenced practice patterns, as well as the generalizability of this data to the current knowledge and physician's adherence to adopt contemporary treatment options which have been integrated within standard treatment algorithms.

Demographic characteristics of metastatic breast cancer patients, diagnosis of disease and treatments initiated for all patients receiving first line (1L) and second line (2L) treatment who were admitted to the clinical centers starting from year 2010 will be retrospectively collected for this study. Data of patients who previously consented for institutional data sharing will be retrieved from patient charts and recorded in a secure electronic registry.

The study data will be categorized on two different patient characteristics: Metastatic pattern at presentation [recurrent metastatic breast cancer (rMBC) or de-novo metastatic breast cancer (dnMBC)] of patient and date of initial presentation for diagnosis and treatment. The study is planning to analyze patients with follow-up data of minimum 3 years and the data recording will eventually plan to construct two cohorts based on the initial diagnosis date; patient diagnosed during Jan 2010-Dec 2014 and Jan 2015-Dec 2019.

The main goal of the study is to define whether if any changes in the treatment practices occurred during the period of data record in line changes occurred with the availability of novel diagnostic methods and treatments for metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no upper age limit.
* Must have a definite diagnosis of metastatic breast cancer at the time of initial application at any of the participating clinical centers.
* Patients who were initiated their first treatment at the center where the initial mBC diagnosis was made and whose follow-up and treatment period have continued at the current center.
* Patients must have signed an informed consent that allow collection of personal data and protection of patient confidentiality according to the standard procedures of each participating center.

Exclusion Criteria:

* Patients who were referred to the participating centers for further treatment for a second opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic breast cancer during January 2010-December 2014 and January 2015-December 2019 who were previously treated at the selected/participating clinical centers.
Sampling Method: Probability Sample
Enrollment: 1331 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Treatment outcome data: Overall survival (OS) | Up to 10 years
  OS: it is defined as the time from the date of initial breast cancer diagnosis to the date of death due to any cause.
  OS data: number (%) patients receiving first-line, second-line, third-line chemotherapy
Treatment outcome data: Progression-free survival (PFS) | Up to 10 years
  PFS: it is defined as the time from the start date of a specific treatment to the documentation of disease progression on such treatment, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
  PFS data: number (%) patients receiving first-line, second-line, third-line chemotherapy

SECONDARY OUTCOMES:
Time to progression (TTP) | Up to 10 years
  Time to progression is measured as the time from study entry to the development of disease progression.
Demographic characteristics at baseline | Up to 10 years
  * Patient demographics: age and gender.
  * Type of insurance (social security system, private insurance) [if available]
Clinical and pathological characteristics: Diagnosis | Up to 10 years
  Date and stage of diagnosis
Clinical and pathological characteristics: Clinical and/or pathological stage | Up to 10 years
  Tumor clinical and/or pathological stage will be collected through the tumor-node-metastasis (TNM) staging system
Clinical and pathological characteristics: Lymph nodes | Up to 10 years
  Number (N) of lymph nodes involved / retrieved
Clinical and pathological characteristics: Tumor size | Up to 10 years
  Measured by a pathologist from the tumor surgical specimen at breast surgery [unifocal, multifocal, multicentric]
Clinical and pathological characteristics: Pathological subtype | Up to 10 years
  Number of patients with different pathological subtypes [HER2+/HR- , HER2+/HR+, HER2-/HR+, TNBC]
Clinical and pathological characteristics: Hormone-receptor expression | Up to 10 years
  Estrogen Receptor positivity [%] Progesterone Receptor positivity [%]
Clinical and pathological characteristics: Human Epidermal Growth Factor Receptor 2 (HER-2) expression | Up to 10 years
  HER2 status will be determined by immunohistochemistry (IHC) [scoring: 0, 1+, 2+, 3+] In situ hybridization (ISH) will be used to confirm IHC results [positive/negative and amplification ratio (%)] Progesteron Receptor positivity [%]
Clinical and pathological characteristics: Histological type | Up to 10 years
  Histological type: Invasive ductal, invasive lobular, other.
Clinical and pathological characteristics: Histological grade | Up to 10 years
  Histological grade with using Modified Bloom Richardson grading system: Grade 1, Grade 2, Grade 3
Clinical and pathological characteristics: Nuclear grade | Up to 10 years
  Nuclear grade: Grade 1, Grade 2, Grade 3
Anatomopathological characteristics of the tumor: Ki-67 | Up to 10 years
  Tumor Ki-67 proliferation index will be collected
Treatment data: type of chemotherapy | Up to 10 years
  Number (%) patients receiving neoadjuvant or adjuvant chemotherapy
Treatment data: adjuvant hormonotherapy | Up to 10 years
  Number (%) patients receiving adjuvant hormonotherapy
Treatment data: radiotherapy | Up to 10 years
  Number (%) patients receiving radiotherapy [Stereotactic Body Radiation Therapy (SBRT), conventional radiotherapy or other]
Treatment data: surgery | Up to 10 years
  Number (%) patients underwent surgery [by regions]
Treatment data: locally ablative treatment | Up to 10 years
  Number (%) patients had locally ablative treatment [by regions]
Follow-up data: initial recurrence | Up to 10 years
  Date and site of recurrence [visceral, non-visceral, central nervous system (CNS) and oligometastatic]
Follow-up data: current condition | Up to 10 years
  The date of the last review and current clinical condition will be recorded.
Follow-up data: date and cause of death | Up to 10 years
  Date and cause of death, when applicable.

CONTACTS AND LOCATIONS:
Locations (6):
- Turkey (Türkiye) (6):
  - Ege University Hospital, Izmir, Bornova
  - Istanbul University, Istanbul, Fatih
  - Acibadem Maslak Hospital, Istanbul, Maslak
  - Marmara University Pendik Training and Research Hospital, Istanbul, Pendik
  - Acibadem Altunizade Hospital, Istanbul, Istanbul, Üsküdar
  - American Hospital, Istanbul, Şişli